CLINICAL TRIAL: NCT05605431
Title: Predictors of Obstructive Sleep Apnea in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Predictors of OSA in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Ibrahim Hassan, Assistant Professor of pulmonology, Cairo University
Other Study IDs: MS-81-2020
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: OSA; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD associated with OSA
  Interventions: Diagnostic Test: Polysomnography
- COPD without OSA
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — over nightSleep study

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea(OSA) are common disorders ,the co-existence of both conditions is called overlap syndrome Smoking , obesity , airway resistance and inflammation are considered risk factors for both conditions ,interestingly either COPD and OSA are associated with increased cardiovascular complications with further increased risk in overlap syndrome Multiple theories could explain that one disorder can predispose or exaggerate the other. For example, in COPD cigarette smoking and inhaled steroids are linked to myopathy of upper airway dilator muscles. Moreover in core-pulmonale redistribution of edema fluid in supine position during sleep can also contribute to or exacerbate OSA .

On the other hand , OSA patients might smoke frequently and more heavily to compensate for excessive daytime sleepiness and to help them to lose weight , which results in exaggerated airway inflammation and exacerbate COPD. Rationale of the study was to assess the prevalence and predictors of OSA among patients with stable COPD.

ELIGIBILITY:
Inclusion Criteria:

* All stable COPD patients

Exclusion Criteria:

* Patients with end organ failure

Ages: 25 Years to 76 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: two groups , COPD with OAS ( OVERLAP SYNDROME) COPD without OSA
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
screening for OSA among COPD | 6 months
  to assess the percentage of OSA among COPD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No